CLINICAL TRIAL: NCT01636492
Title: Single Oral Ascending Dose Study of Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of RO4917838 in Healthy Male Volunteers.
Brief Title: A Study of Bitopertin (RO4917838) in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: BP19292
Record Dates: First submitted 2012-07-06; First posted 2012-07-10 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — (4-(3-fluoro-5-trifluoromethylpyridin-2-yl)piperazin-1-yl)(5-methanesulfonyl-2-(2,2,2-trifluoro-1-methylethoxy)phenyl)methanone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Bitopertin (Experimental)
  Interventions: Drug: bitopertin
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: bitopertin — Single oral dose
  Arms: Bitopertin
Drug: placebo — Single oral dose
  Arms: Placebo

SUMMARY:
This randomized, double-blind, placebo-controlled, dose-escalating study will evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of bitopertin in healthy male volunteers. Subjects will be randomized in cohorts to receive single oral doses of either bitopertin or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male healthy volunteer, 18 to 60 years of age inclusive
* Body mass index (BMI) 19-35 kg/m2 inclusive
* Supine blood pressure within the normal range of the center and heart rate >/= 40 provided QTcB is <450 ms
* Subjects must agree to use a barrier method of contraception (e.g. condom) for the duration of the study and for 30 days after study completion

Exclusion Criteria:

* History or evidence of any clinically significant disease or disorder
* Clinically significant ECG abnormalities
* Positive for hepatitis B, hepatitis C or HIV infection
* Previous treatment with iron for iron deficiency anemia
* Regular smoker (>10 cigarettes, >3 pipefuls or >3 cigars per day)
* History of alcohol and/or drug abuse or addiction within the last 2 years before study start
* Any confirmed significant allergic reactions against any drug, or multiple allergies in the judgment of the investigator
* Participation in a clinical study with an investigational drug within the last three months prior to screening
* Any condition or disease detected during the medical interview/physical examination that would render the subject unsuitable for the study, place the subject at undue risk or interfere with the ability of the subject to complete the study in the opinion of the investigators or their designee

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2005-11; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | 17 days

SECONDARY OUTCOMES:
Pharmacokinetics: Area under the concentration-time curve | Pre-dose and 1, 2, 4, 8, 12, 24, 72, 96, 144, 168 (+/-8), 216 (+/-24), 288 (1/-48) hours post-dose
Pharmacokinetics: Urine concentrations drug/metabolites | Pre-dose and up to 72 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Christchurch, New Zealand